CLINICAL TRIAL: NCT07121127
Title: Effect of Fu's Subcutaneous Needling for Age-related Macular Degeneration
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhiming Yan (Other)
Responsible Party: Sponsor-Investigator, Zhiming Yan, postgraduate of the Second Clinical College of Guangzhou University of Chinese Medicine, Guangdong Provincial Hospital of Traditional Chinese Medicine
Organization: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZF2025-237-01
Record Dates: First submitted 2025-08-01; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Age - Related Macular Degeneration (AMD)
Keywords: Fu's subcutaneous needling; age-related macular degeneration; OCTA
MeSH Terms: conditions — Macular Degeneration | interventions — Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fu's subcutaneous needling group (Experimental): Fu's subcutaneous needling group with oral Vitamin C and vitamin E supplements
  Interventions: Combination Product: FSN+Vitamin supplement
- Control group (Other): oral Vitamin C and vitamin E supplements
  Interventions: Drug: Vitamin Supplements

INTERVENTIONS:
Combination Product: FSN+Vitamin supplement — Fu's subcutaneous needling with oral Vitamin C and vitamin E supplements
  Arms: Fu's subcutaneous needling group
Drug: Vitamin Supplements — oral Vitamin C and vitamin E supplements
  Arms: Control group

SUMMARY:
This pilot randomized controlled trial aims to evaluate the efficacy and safety of FSN in improving symptoms in patients with dAMD.38 eligible participants will be recruited and randomly assign them in a 1:1 ratio to the FSN group and the control group. Throughout the study, both groups will take oral vitamin C and vitamin E supplements for a total of 28 days. Participants in the FSN group will receive four treatment sessions over two weeks. Both groups will be assessed at the end of the FSN treating period during the mid-study period, with ocular blood flow dynamics measured using OCTA, followed by a two-week follow-up. The primary outcome of this trial is the change in visual acuity from baseline to week 2, with secondary outcomes including visual field, visual function scale, macular thickness, central avascular zone area vascular density, and choroidal thickness.

ELIGIBILITY:
Inclusion Criteria:

（ 1 ） Age between 50 and 85 years old with no gender restrictions （ 2 ） Meets the diagnostic criteria for dry age-related macular degeneration (AMD) as outlined in the 2023 Chinese Clinical Practice Guidelines for Age-Related Macular Degeneration （ 3 ） Both monocular and binocular cases of dry AMD are included. For patients with bilateral lesions the experimental group is based on the patient's preferred eye (if both eyes are preferred the average of the data collected from both eyes is included in the analysis) （ 4 ） Participants must voluntarily consent and sign an informed consent form and be willing to cooperate with follow-up visits.

Exclusion Criteria:

（ 1 ） Serious eye diseases that significantly affect the condition of the fundus excluding dry macular degeneration including fundus lesions such as fundus hemorrhage and wet macular degeneration; or concomitant eye diseases requiring immediate treatment such as acute glaucoma; severe opacity of the refractive media such as mature cataracts （ 2 ） In distance vision testing the patient cannot discern the direction of the largest character at a distance of 1 meter from the distance vision chart （ 3 ） Participants who have undergone eye surgery within the past six months （ 4 ） Participants with non-ophthalmic conditions that may severely affect vision such as large-area cerebral infarction cerebral hemorrhage diabetes thyroid eye disease vitamin A deficiency or Sjögren's syndrome （ 5 ） Pregnant or lactating women （ 6 ） Participants with severe anemia renal failure acute phase of cardiovascular disease implanted cardiac pacemaker thrombocytopenia or other hematological conditions with a high risk of severe subcutaneous bleeding or requiring skin puncture （ 7 ） Participants who have taken medications or consumed foods that affect ocular blood supply within the past week such as caffeine atropine or other treatments for macular degeneration （ 8 ） Participants who require contact lenses.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-07-07 (Estimated); Primary Completion 2029-08-08 (Estimated); Study Completion 2030-03-09 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | Day 14
  The best corrected visual acuity at distance and near will be tested as the main outcome after 2-week treatment，which is the mid period of intervention.During vision testing, paticipants stand 5 meters from the chart with one eye covered. The chart height is adjusted so the 1.0 line aligns with their eye level. For near vision assessment, the subject positions themselves 25 cm from the vision chart with one eye occluded.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity | FSN group:Baseline 2 days in FSN treatment period(days 4 and 11),follow-up day (day 28);Control group: Baseline follow-up day (day 28)
  Measuring vision at different time points compared with the primary outcome
Visual Function Questionnaire 25 | both groups:baseline, end of FSN treatment week (day 14) follow-up day (day 28)
  The NEI-VFQ-25 is a 25-item version questionnaire of the NEI-VFQ (National Eye Institute Visual Functioning Questionnaire),widely applied in ophthalmic studies including cataract and macular degeneration, with established reliability and validity. The Chinese version was created through cultural adaptation and professional translation. This study employs the version provided by Zhongshan Ophthalmic Center, Sun Yat-sen University.The questionnaire comprises two subscales: visual function (12 items) and quality of life (13 items). Each item scores from 0(worst) to 100(best) , where higher scores indicate better quality of life. Different from the English original's 5/6-point scale, the Chinese version converted to 4 point scale scoring follows a reverse-calculation method: each question's score equals 4 points minus the points selected. Domain scores are summed to generate the total visual function score.
OCTA metrics | baseline ,end of the FSN treatment week (day 14)
  The SPECTRALIS OCT Angiography Module (Heidelberg Engineering) was utilized for fundus blood flow signal acquisition. FAZ,VD,CMT and CT will be collected as OCTA metrics of dAMD.The"FAZ Measurement" function will automatically quantify the foveal avascular zone (FAZ) area (mm²), corresponding to the superficial capillary plexus (SCP) of the macula ,and the "Density"function quantifies vessel density (VD) and automatically generates an en face projection map, providing the percentage of vascular area occupancy across the entire macula, with regional analyses of the fovea, parafovea, and temporal/superior/nasal/inferior macular sectors.The digital calipers tool within the OCT software was utilized to measure central foveal thickness (CFT) and central macular thickness (CMT).Choroid thickness (CT) will be measured vertical distance from the outer edge of the retinal pigment epithelium to the choroidal-scleral interface manually.
Visual field | both groups:baseline, end of FSN treatment week (day 14) follow-up day (day 28)
  The Humphrey Field Analyzer enables precise quantitative measurement of retinal light sensitivity thresholds with SITA Standard program 10-2, specifically applicable for macular field testing.Operators perform visual field examinations via touchscreen or keyboard interface at pre-treatment, post-treatment, and follow-up phases. During testing, the patient remains seated with the non-tested eye occluded, stabilizes their chin and fixates on the central target of the gaze tracking system. Each perceived light stimulus triggers a press of the handheld response button. If patients feel tired, a prolonged button press can activate a pause, allowing them to rest before resuming the measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Sun, Principal Investigator — Guangzhou University of Chinese Medicine - Department of Acupuncture and Rehabilitation Clinical Medicine

IPD SHARING:
Plan to Share IPD: Yes
Paper publication or Resman
Supporting Information: Study Protocol, SAP, ICF, CSR